CLINICAL TRIAL: NCT07327606
Title: A Prospective Cohort Study on Prognostic Factors in Patients With Cardiovascular-kidney-metabolic Syndrome
Status: Recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M20250184
Record Dates: First submitted 2025-12-26; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-03

CONDITIONS: Patient With Cardiovascular-kidney-metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months

SUMMARY:
Patients with Cardiovascular-kidney-metabolic syndrome (CKM) will be prospectively enrolled. We will conduct comprehensive analyses, including transcriptomics, proteomics, and metabolomics, using various types of samples such as plasma and whole blood. Adenosine stress echocardiography will be monitored to collect a large amount of data. Long-term follow-up will be conducted, and modern information technology will be utilized to analyze the relationship between different biomarkers and prognosis. Combined with clinical data, we will attempt to construct a predictive model for CKM patients to precisely formulate treatment and follow-up strategies. Demographic and basic clinical information of the study subjects will be collected, including age, gender, height, weight, blood pressure, cardiovascular risk factors (smoking history, alcohol consumption history, blood pressure, lipid levels, glycated hemoglobin, fasting blood glucose, etc.), clinical medication use, and coronary angiography images. During follow-up, changes in risk factor-related indicators such as blood pressure, blood glucose, and lipid levels, medication use, inflammatory markers, and stress echocardiography will be recorded. Plasma and whole blood samples will be collected and stored in a biobank managed by a biospecimen management system. The occurrence of major adverse cardiovascular events (MACE) in all enrolled patients during the follow-up period will be statistically analyzed. This cohort study will follow up with patients for at least 3 years using multiple methods (questionnaires, outpatient follow-up, and telephone calls). Changes in indicators such as MACE occurrence, biochemical markers, echocardiography, carotid ultrasound, and stress echocardiography will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* 1）Patients who meet the criteria for CKM stages 0-4 were included. 2）Clinical data were complete.

Exclusion Criteria:

* 1) Presence of infectious diseases during the sample retention period. 2) Presence of autoimmune diseases, such as systemic lupus erythematosus, rheumatoid arthritis, systemic sclerosis, vasculitis, etc.

  3) Presence of tumors. 4) Patients with an estimated life expectancy of less than 2 years. 5) Patients with known hypersensitivity to adenosine. 6) Patients who cannot follow up regularly. 7) Pregnant or breastfeeding women, and those participating in other clinical trials.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who meet the criteria for Cardiovascular-kidney-metabolic syndrome. Stage 1: Excess or abnormal fat accumulation, such as overweight/obesity, abdominal obesity, or normal function of adipose tissue, without other metabolic risk factors or CKD.
  Stage 2: Presence of metabolic risk factors and CKD, such as having metabolic risk factors (hypertriglyceridemia ≥135 mg/dL, hypertension, diabetes, metabolic syndrome) or moderate to high-risk CKD.
  Stage 3: Presence of CKM with subclinical CVD, or being at an equivalent level of risk (assessed as high-risk CVD or very high-risk CKD).
  Stage 4: Presence of CKM with CVD, with Stage 4a without renal failure; Stage 4b with renal failure.
Sampling Method: Non-Probability Sample
Enrollment: 4526 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular event | 3 years
  Cardiovascular death, non-fatal myocardial infarction, non-fatal stroke, and revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Ming Cui, Study Director — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China